CLINICAL TRIAL: NCT06174246
Title: Optimization of a Chronic Pain Self-management Program - a Pilot Randomized Clinical Trial
Brief Title: Pain Education Program Optimization (PEPO) Trial
Acronym: PEPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Quebec Pain Research Network (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-2935
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: Randomized Controlled Trial; Patient Education as Topic; Self-Management; Non-Cancer Chronic Pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: Self-management program, with or without support from a physiotherapist.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment is masked as all outcomes are derived from self-administered questionnaires that will be filled online without the presence of any member of the research team.
  Data analysis will be masked (intervention groups will be coded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain self-management (Active Comparator): Participants will complete an online pain self-management education program by themselves as it is intended.
  Interventions: Behavioral: Pain self-management program
- Pain self-management with support from a physiotherapist (Experimental): Participants will complete an online pain self-management education program, and, during the treatment period, will take part in two sessions with a physiotherapist and one group session led by a peer living with chronic MSKP.
  Interventions: Behavioral: Pain self-management program; Behavioral: Additional support for self-management program

INTERVENTIONS:
Behavioral: Pain self-management program — Agir pour moi (Acting for me) is a chronic pain self-management program designed to be followed independently online. The eight modules, normally spread over eight weeks and taking about 60 to 90 minutes per week to complete, focus on different strategies for managing pain on a daily basis.
  The structured lessons include videos, audio capsules, activities, and written information, also provided in an audio format. The program covers goal setting, stress management through relaxation, breathing and mindfulness, pacing, physical activity, thoughts and emotions, sleep, nutrition, flare-up management, and planning.
  The program was developed through a partnership between various chronic pain interest groups, and is hosted and managed by the Leadership Chair in Chronic Pain Education.-MEDISCA de l'Université Laval, Québec, Canada.
  See ClinicalTrials entry NCT05319652 https://gerermadouleur.ca/agir-pour-moi/
  Other Names: "Agir pour moi" (Acting for me)
Behavioral: Additional support for self-management program — This intervention is designed to give extra support to patients completing the online pain education program. It consists of two visits with a physiotherapist, and one group session led by a peer living with chronic musculoskeletal pain.
  Sessions with the physiotherapist will occur at the beginning of the program and at the midway point. They will be used first to present the objectives and the components of the self-management program, to reinforce its potential to improve the participant's ability to manage their pain, and then to answer the participant's questions on the program and follow up on the regular completion of the lessons.
  The group session will be co-facilitated by a physiotherapist and a patient-partner, and will include participants who have completed at least six weeks of the program. It will serve as a discussion forum to share helpful pain self-management strategies, lived experiences with pain and facilitators in completing the program.
  Arms: Pain self-management with support from a physiotherapist

SUMMARY:
The goal of this clinical trial is to compare two different modes of delivering a self-management program for chronic pain (independently vs. with additional support) on pain-related disability.

Participants with chronic musculoskeletal pain will take part in a 10-week online pain self-management program. For the participants in the group with additional support, the intervention will also include two physiotherapist-led sessions and one group session with other participants.

The hypothesis is that the results will support that both modes of delivery could be effective, but the self-management program with additional support will be more effective for reducing pain intensity and pain disability compared to the self-management program alone.

DETAILED DESCRIPTION:
The primary objective of this pilot randomized controlled trial (RCT) is to compare the short-, mid-, and long-term effects (10 and 26 weeks following the start of the intervention) of two different modes of delivering a self-management program for chronic pain (self-management vs. enhanced self-management, offering two physiotherapist-led and one patient-partner-led sessions) on pain-related disability in a group of patients with chronic musculoskeletal (MSK) pain. Secondary objectives include comparing the effects of the two delivery modes on pain severity and on psychological constructs related to pain, namely kinesiophobia, catastrophizing, pain self-efficacy, anxiety, and depression.

The hypothesis is that the results will support both modes of delivery, but that the enhanced self-management program will lead to larger effects on pain-related disability and pain intensity.

Methodology Participants: 86 adults (aged between 18 and 75) with chronic MSK pain (>3 months) will be included. Potential participants will be recruited from waiting lists of pain-management programs and through email lists and social media.

Study design: This parallel group RCT will include three evaluation sessions over six months (baseline, 10 and 26 weeks) and, for the enhanced self-management group, three in-person meetings over 10 weeks. Questionnaires will be completed online using the REDCap web application. At baseline, participants will first complete a questionnaire on sociodemographic, symptomatology and comorbidity. Self-administered questionnaires for assessing primary and secondary outcomes will be completed by participants at all evaluation sessions. A global rating of change question will also be completed at 10 and 26 weeks. For the enhanced self-management group, the in-person meetings will be carried out at Centre interdisciplinaire de recherche en réadaptation et intégration sociale (Cirris). Ethics approval has been obtained from the sectorial rehabilitation and social integration research ethics committee of the CIUSSS-CN (project #2024-2935).

Randomisation/blinding: A randomisation list has established prior to the beginning of the study using a random number generator. An independent research assistant not involved in data collection generated the randomisation list. Randomisation is stratified to ensure balance of the treatment groups with respect to self-reported gender (3 categories : man, woman, and all other gender identities). A blocked randomisation was used to make sure that two equal groups of 43 participants will be obtained. Participants will be unaware of the intervention delivery mode received by the other group.

Outcomes: Outcomes were selected based on Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) recommendations, which attest to the good psychometric properties of the selected outcomes. See the outcomes section for details on primary and secondary outcomes measures.

Statistical analyses: Descriptive statistics will be used for all outcome measures at each measurement time to summarise results. The dataset will also be explored to check the distribution of the data. The effect sizes (Cohen's d) will be calculated between groups at each timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Having musculoskeletal pain for more than 3 months.

Exclusion Criteria:

* Unable to participate throughout the 26 weeks of the study.
* Having a diagnosis of rheumatoid, inflammatory or neurodegenerative diseases, fibromyalgia or of complex regional pain syndrome.
* Having received a corticosteroid injection in the previous twelve weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain-related functional limitations | Change from baseline at 10 weeks, change from baseline at 26 weeks
  The Pain Interference subscale from the short-form of the Brief Pain Inventory questionnaire (BPI-SF).
  Calculated as the mean of the seven interferences items of the BPI-SF, with a score ranging from 0 (does not interfere) to 10 (completely interferes).

SECONDARY OUTCOMES:
Pain Severity | Change from baseline at 10 weeks, change from baseline at 26 weeks
  The Pain Severity subscale from the short form of the Brief Pain Inventory questionnaire (BPI-SF).
  Calculated as the mean of the four items on pain severity of the BPI-SF, with a score ranging from 0 (No pain) to 10 (Pain as bad as you can imagine).
Kinesiophobia | Change from baseline at 10 weeks, change from baseline at 26 weeks
  The 13-item Tampa Scale of Kinesiophobia (TSK-13). Each item is scored on a 1 to 4 scale, with a total score ranging from 13 (least kinesiophobia) to 52 (most kinesiophobia).
Pain catastrophizing | Change from baseline at 10 weeks, change from baseline at 26 weeks
  The 6-item short form of the Pain Catastrophizing Scale (PCS-6). Calculated as the sum of the 6 items, with a score ranging from 0 (lowest level of pain catastrophizing) to 24 (highest level of pain catastrophizing).
Pain-related Self-Efficacy | Change from baseline at 10 weeks, change from baseline at 26 weeks
  The 10-item Pain Self-Efficacy Questionnaire (PSEQ-10). Score ranges from 0 to 60, where high scores indicate greater levels of confidence in dealing with pain.
Anxiety and Depression | Change from baseline at 10 weeks, change from baseline at 26 weeks
  The 4-item Patient Health Questionnaire (PHQ-4). Calculated as the sum of the 4 items, with a score ranging from 0 (no signs or symptoms) to 12 (most severe signs and symptoms).
Patient Acceptable Symptom State (PASS) | At baseline, 10 weeks, and 26 weeks
  PASS simple question ("Taking into account all your activities of daily living, your level of pain, and also your functional limitations, do you consider your current condition to be satisfactory?"), answered by "Yes" or "No".
Global condition change since start of intervention, assessed by a global rating of change question | At 10 weeks and 26 weeks
  A global rating of change question ("Overall, have you noticed any change in your condition since you entered the research project [start of intervention]?"), answered on a 15-item Likert scale ranging from -7 (Very greatly deteriorated) to 7 (Very greatly improved).
Patient satisfaction with intervention | At 10 weeks (end of intervention period)
  4 questions to ask the participants if they are satisfied of :
  1. the intervention they received globally;
  2. the intervention mode, i.e. the way it was delivered;
  3. the content of the sessions;
  4. the tools they received to apply the advice received. The choice of answers for each question is : "Unsatisfied" or "Satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, PhD, Principal Investigator — Laval University
Locations (1):
- Cirris (Centre interdisciplinaire de recherche en réadaptation et intégration sociale), Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the self-management pain education program, hosted and managed by the Quebec Pain Research Network (QPRN). — https://gerermadouleur.ca/en/